CLINICAL TRIAL: NCT01757587
Title: Evaluation of Galvus (Vildagliptin) Efficacy Versus Placebo in Patients With Type 2 Diabetes, Inadequately Controlled by Metformin and Basal Insulin, This One Having Been Properly Titrated.
Brief Title: Galvus (Vildagliptin) vs Placebo in Combination With Metformin and Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-001813-14
Record Dates: First submitted 2012-02-08; First posted 2012-12-31 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Galvus; basal insulin; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin (Active Comparator)
  Interventions: Drug: Vildagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin — 50 mg, 2 tablets/day on 3 months, both periods of treatment
  Other Names: Metformin and basal insulin
  Arms: Vildagliptin
Drug: Placebo — 50mg 2 tablets / day on 3 months, both periods of treatment
  Other Names: Metformin and insulin basal
  Arms: Placebo

SUMMARY:
The main objective is to show that the addition of Galvus versus placebo in patients with type 2 diabetes treated with metformin (at the maximum tolerated dose) and basal insulin properly titrated, allows a greater proportion of patients achieving an HbA1c below 7%.

The primary efficacy endpoint was the percentage of patients responding to treatment (HbA1c less than 7%) after 3 months of treatment with Galvus or placebo

DETAILED DESCRIPTION:
* Visit V1 : screening
* Inclusion visit V2: Be verified inclusion criteria of patient. At the inclusion visit will be collected:

  * Informed consent to participate in the study…
  * The following data: age, duration of diabetes, usual basal insulin dose, other co-morbidities : hypertension, complications of diabetes, dyslipidemia, smoking (and their associated treatments).
  * Data from physical examination and in particular: weight, BMI, waist circumference, systolic blood pressure (SBP) and diastolic (DBP)
  * Therapeutic adjustments can be made. In the case of inefficient combination with a sulphonylurea (HbA1c> 7%), it will be stopped and basal insulin will be titrated during the run- in period (2 months) in order to obtain a good control of fasting glucose.
* Visit V3 : At the randomization visit, be collected the results of HbA1c and other biological assessment (FPG, fasting lipid profile). Moreover, the insulin will be collected and the patient will receive the treatment for 3 months (for ex Galvus in this case according to randomisation).
* Visit V4a the glycemic holter will be introduced and removed 5 days later (at visit V4B). The interstitial glucose will be calibrated during the Holter by the blood glucose. When collecting the glycemic holter, patients will also have a clinical examination and a new biological assessment (HbA1c, FPG, C peptide, fasting lipids ...) and an assessment of their dietary intake during the port the holter (overall calorie intake: cal + G, L, P)
* Visit V5 : the patient will receive the treatment for 3 months (placebo at this visit according the example cited above ).
* Visit V6A, it will be the same as for the visit V4a, the glycemic holter will be introduced and removed at V6B visit. Similarly, in the collection of glycemic holter, patients will also have a new clinical examination, laboratory evaluation (HbA1c, FPG, fasting lipids ...) and a dietary assessment (overall calorie intake: cal + G, L, P).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for at least 3 months with metformin (at the maximum tolerated dose (for at least 1 month) + / - sulfamide and basal insulin
* Patient with an HbA1c between 7 and 9% at the inclusion visit
* Patients able to use a continuous glucose monitoring system,

Exclusion Criteria:

* Patients already receiving a specific treatment of postprandial (GLP1, ..)
* Patients with type 1 diabetes, or secondary diabetes
* Patients with eating disorders
* Patients with major complications of diabetes
* Patients participating in another clinical trial
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients responding to treatment (HbA1c less than 7%) | after 3 months of treatment with Galvus or placebo

SECONDARY OUTCOMES:
Compare HbA1c and other clinical and laboratory parameters (fasting plasma glucose (FPG), fasting lipids, weight) | after 3 months of treatment with Galvus or placebo

OTHER OUTCOMES:
Evaluate more precisely the optimized glycemic control through a glycemic holter | after 3 months of treatment with Galvus or placebo
  Safety criteria: number of symptomatic hypoglycemia episodes and number of severe hypoglycemic events

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia FRANC, MD, Principal Investigator — CH Sud Francilien
Locations (1):
- CH Sud Francilien, Évry, France